CLINICAL TRIAL: NCT04691076
Title: Efficacy and Safety of Low-dose Esketamine Combined With Target-controlled Infusion of Propofol for Painless Gastrointestinal Endoscopy and Polypectomy
Brief Title: Effect of Low-dose Esketamine Combined With Target-controlled Infusion of Propofol for Painless Gastrointestinal Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Union Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TYang001
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Pain; Anesthesia
Keywords: Esketamine; Gastrointestinal endoscopy; Analgesia; Sedation; Respiratory depression
MeSH Terms: conditions — Pain; Agnosia; Respiratory Insufficiency | interventions — Propofol; Esketamine; Fentanyl

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol/Esketamine sedation (Experimental): Propofol target-controlled infusion is performed first,when the infusion concentration reaches 1.5μg/ml,esketamine 0.15mg/kg is injected intravenously;then the dose is adjusted according to the depth of anesthesia and the modified observer's assessment of alert /sedation scale, and propofol target-controlled infusion for every increase of 5μg/ml in concentration, the corresponding increase of esketamine is 0.05mg/kg; the total dose of esketamine used in surgery shall not exceed 0.5mg/kg.
  Interventions: Drug: Propofol; Drug: Esketamine
- Propofol/Fentanyl sedation (Active Comparator): Propofol target-controlled infusion is performed first.When the infusion concentration reaches 1.5μg/ml, fentanyl 0.6μg/kg is injected intravenously; then the dose is adjusted according to the depth of anesthesia and the modified observer's assessment of alert /sedation scale, and propofol target-controlled infusion for every increase of 5μg/ml in concentration,the corresponding increase of fentanyl is 0.2ug/kg; the total dose of fentanyl used in surgery shall not exceed 1.2ug/kg.
  Interventions: Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — Propofol is administered by target-controlled infusion
Drug: Esketamine — Esketamine is intravenously administrated
  Arms: Propofol/Esketamine sedation
Drug: Fentanyl — Fentanyl is intravenously administrated
  Arms: Propofol/Fentanyl sedation

SUMMARY:
Purpose: 1. To determine the efficacy of low-dose esketamine in painless gastrointestinal endoscopy. 2. To determine the safety of low-dose esketamine in painless gastrointestinal endoscopy. 3. To provide a theoretical basis and new ideas for the application of esketamine as a new drug in perioperative period.

DETAILED DESCRIPTION:
Keeping spontaneous breathing anesthesia can provide patients with comfortable diagnosis and treatment experience during gastrointestinal endoscopy, which is a vital prerequisite for the large-scale development of this operation as well as the early screening and treatment of gastrointestinal malignancies. Clinically, fentanyl combined with propofol is the most commonly used anesthesia regimen for the painless gastroscopy, however its high incidence of respiratory and circulatory depression will threaten the safety of patients. Instead, esketamine has a good action in anesthesia and analgesics, a slighter respiratory depression, as well as with a remarkable improvement in adverse effects than ketamine. What has already been proved is that low- dose of esketamine can remarkably reduce the dosage of propofol during endoscopic retrograde cholangiopancreatography; In our pilot study, we found that not only the incidence of respiratory depression was significantly lower than that of fentanyl during endoscopic polypectomy, but also the dosage of propofol was reduced at the same time,suggesting that esketamine may have a potential superiority in the painless gastrointestinal endoscopy.Our project plans to collect the patients who have received painless gastroscopy and polypectomy in the hospital, and use a target-controlled infusion (TCI) of propofol in combination with esketamine, by observing the total dose of propofol , the time of recovery and the length of hospital stay, the satisfaction of patients and endoscopists, drug side effects,adverse events of respiratory and circulatory system and other indicators ,to evaluate the efficacy and safety of this anesthetic scheme.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's American Society of Anesthesiologists physical status is I-III.
2. Subject has no symptoms of allergy to anesthetics.
3. Subject has no contraindications for gastrointestinal endoscopy.
4. Subject has given written informed consent to participate.

Exclusion Criteria:

1. Subject's BMI <18 or >30
2. Subject has poorly controlled or untreated hypertension.
3. Subject has severe ischemic heart disease.
4. Subject is an untreated or undertreated patient with hyperthyroidism.
5. Subject has used drugs that affect their central nervous system.
6. .Subject has mental illness.
7. .Subject has epilepsy.
8. .Subject has a history of chronic pain.
9. .Subject is pregnant or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative propofol Consumption | intraoperative
  Total amount of propofol administered intraoperatively

SECONDARY OUTCOMES:
The incidence of adverse events in pulmonary and circulatory systems | During the operation
  Pulmonary incidents include:Decreased blood oxygen saturation (SpO2 drops to 75%~90%, duration <60s);Severe decrease in blood oxygen saturation (SpO2<90%, duration>60s; or SpO2<75%);Obstruction of the airways occurs and requires the use of jaw manipulation or emergency airway equipment.
  Cardiovascular incidents include:
  Bradycardia or tachycardia; Arterial blood pressure increased or decreased by more than 20% of the baseline; Other matters requiring urgent attention.
Time of recovery, post-anaesthesia care unit and discharge from hospital | procedure ( the end of endoscopy removal)
  When the patient is successfully resuscitated,record the time in post-anaesthesia care unit and the time when the discharge standards are met.
The incidence of side effects of esketamine | Intraoperative
  Record the adverse effects of esketamine such as dizziness, nausea, etc.
The number of patients'body movement during operation | During the operation
  Record the patient's body movement during the operation, which reflects the level of sedation.
The satisfaction of the endoscopist and patient | 24 hours after surgery
  Patients fill out questionnaires before and after surgery to record pain, sedation levels, and side effects (such as nausea and dizziness) to assess their satisfaction,meanwhile,telephone calls can be made one day after the surgery to evaluate their postoperative satisfaction.In addition, the satisfaction of the endoscopist with the sedation level could also recorded on a questionnaire after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, Principal Investigator — Tianjin Union Medical Center
Locations (1):
- Tianjin Union Medical Center, Tianjin, China